CLINICAL TRIAL: NCT06847802
Title: Delphi Process to Achieve Global Consensus on Gender Equity in Critical Care
Status: Not yet recruiting | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Sheila Nainan Myatra, Professor, Dept of Anaesthesia, Tata Memorial Centre
Other Study IDs: 2102
Record Dates: First submitted 2025-02-18; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Professional Role; Research Peer Review
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — The survey will include statements related to the Domains Addressing healthcare workers/trainees, Critical Care (CC) Academic meetings, At the Workplace, CC Academia, Education of CC Trainees, Professionalism and Misconduct, Administration and Governance in the Workplace and in CC Societies, Environmental and logistic facilities, Publication of Gender metrics, Committee/working group for gender-balance The statements related to the domains will be drafted in the form of a 7-point Likert scale (strongly agree, agree, somewhat agree, neither agree nor disagree, somewhat disagree, disagree, strongly disagree) Statements that achieved consensus and stability will be used to issue the position. The results of the Delphi rounds, position statements, and the manuscript will be reviewed and approved by the panelists before submission for publication

SUMMARY:
Gender inequalities in healthcare, including among critical care professionals, have been widely recognized over the last decade. Significant gender disparities persist in areas including leadership, academia, research, workplace remuneration, and medical publication among critical care professionals. Furthermore, there remains a notable gap in knowledge and awareness regarding gender equity (all genders) and inclusivity among healthcare professionals.

Given the limited research and evidence on these issues, Investigator propose employing the Delphi methodology to generate consensus among global critical care practitioners on position statements aimed at addressing gender equity (all genders) in critical care.

DETAILED DESCRIPTION:
To generate consensus among a diverse panel of critical care practitioners, scientists, and researchers on the strategic measures to achieve gender equity in critical care within healthcare institutions, professional societies, organizations, and boards in various professional domains.

ELIGIBILITY:
Inclusion Criteria:

* Professionals working in Intensive Care, Critical Care Practitioner, Scientists, or Researcher
* Any one of the following: having publications, engagement in advocacy related to gender equity, and currently or in the past holding an official leadership position in the Critical Care Society, Intensive care unit, or a healthcare institution
* Completed the Harvard Implicit Association Test (IAT)5

Exclusion Criteria:

* unwilling to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — To achieve gender equity in critical care within healthcare institutions, professional societies, organizations, and boards in various professional domains.
Study Population: Healthy volunteers working in Intensive Care, Critical Care Practitioner, Scientists, or Researcher
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Gender equity among a diverse panel of critical care practitioners, scientists, and researchers in critical care | 1 year
  To generate consensus among a diverse panel of critical care practitioners, scientists, and researchers on the strategic measures to achieve gender equity in critical care within healthcare institutions, professional societies, organizations, and boards in various professional domains.

IPD SHARING:
Plan to Share IPD: No